CLINICAL TRIAL: NCT01143363
Title: Acute Effects of High-intensity Intermittent Sprinting vs. Moderate Intensity Continuous Cycling on Appetite Control on Obese Volunteers
Brief Title: Effect of High-intensity Intermittent Sprinting on Appetite Control on Obese Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Midt-Norge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2010/444-7
Record Dates: First submitted 2010-06-02; First posted 2010-06-14 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
Keywords: Obesity; exercise; appetite; hunger; satiety; food intake
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Resting - control (Placebo Comparator): No exercise
  Interventions: Behavioral: resting - control
- Moderate intensity exercise (Experimental): Moderate intensity exercise (continuous) 1h after breakfast
  Interventions: Behavioral: Moderate intensity exercise
- High intensity intermittent training (Experimental): High intensity intermittent training 1h after breakfast
  Interventions: Behavioral: High intensity intermittent training
- Short sprint (Experimental): Short sprint 1h after breakfast
  Interventions: Behavioral: Short sprint

INTERVENTIONS:
Behavioral: resting - control
  Arms: Resting - control
Behavioral: Moderate intensity exercise
  Arms: Moderate intensity exercise
Behavioral: High intensity intermittent training
  Arms: High intensity intermittent training
Behavioral: Short sprint
  Arms: Short sprint

SUMMARY:
Several studies have shown that high intensity intermittent sprints (HIIS) are more effective than moderate intensity continuous cycling (MICC) in reducing fat mass and improving insulin resistance in normal weight individuals. Changes in the appetite-regulatory system in response to exercise are likely to explain, at least partially, the better outcome observed after HIIS. Unfortunately, there are no studies comparing the impact of different types of acute aerobic exercise on the release of appetite-regulating hormones, subjective feelings of appetite and subsequent energy intake (EI).

The primary objective of this study is to investigate the effects of acute isocaloric bouts of HIIT and MICC or a short duration sprint, in comparison with a resting control condition, on the postprandial release of appetite-regulating hormones, subjective feelings of appetite and subsequent EI in obese individuals. The investigators hypothesize that an isocaloric session of HIIS will result in a better short-term appetite control compared with MICC, by reducing hunger feelings and subsequent food intake more than MICC and by inducing a larger increase in the release of satiety gut peptides compared with the MICC.

DETAILED DESCRIPTION:
This will be a randomised cross-over study with four legs. Participants will act as their own controls and will be assigned to the four experimental conditions (resting, HIIS, MICC and SDS), 1 week apart, in a counter-balanced order.

Participants will be asked to come to the Unit five times: one preliminary session and four experimental conditions (resting, HIIS and MICC isocaloric sessions and SDS). In the preliminary session, anthropometric data (weight and height) will be collected and a maximal fitness test performed, using a cycle ergometer.

For the four experimental conditions, participants will be asked to arrive at approximately 8.00, having fasted for at least 10 hours, and a cannula will be inserted into an antecubital vein. Two fasting blood samples will be taken and a standard breakfast offered. After that, serial blood samples will be taken at regular intervals for a period of 3h.

Participants will be asked to rate their subjective feelings of hunger and fullness using visual analogue scales (VAS) throughout each study morning at different time points. Three hours after breakfast, participants will be placed in individual rooms, presented with a standardized lunch and instructed to rate the taste and palatability of the food presented.

ELIGIBILITY:
Inclusion Criteria:

* an inactive lifestyle,
* weight stable on the previous 3 months,
* not currently dieting to loose weight
* restraint score derived from the Three Factor Eating Behaviour Questionnaire ≤12

Exclusion Criteria:

* history of coronary heart disease,
* type 1 or type 2 diabetes,
* anaemia,
* gout,
* depression or other psychological disorders,
* eating disorders,
* drug or alcohol abuse within the last two years,
* current medication known to affect appetite or induce weight loss and hypertension.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in gut peptides | Blood samples taken in fasting and postprandially for 3h

SECONDARY OUTCOMES:
Food intake at test meal | 3h after breakfast
  Food intake at a test meal will be assessed 3h after breakfast (at 180 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Catia Martins, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Martins C, Stensvold D, Finlayson G, Holst J, Wisloff U, Kulseng B, Morgan L, King NA. Effect of moderate- and high-intensity acute exercise on appetite in obese individuals. Med Sci Sports Exerc. 2015 Jan;47(1):40-8. doi: 10.1249/MSS.0000000000000372. PMID 24824772